CLINICAL TRIAL: NCT06500091
Title: A Multicenter, Open-Label, Single-Arm, Multi-Cohort Phase II Clinical Trial Evaluating the Efficacy and Safety of TQB2916 Injection in Combination With Chemotherapy or in Combination With Penpulimab Injection for Solid Tumors
Brief Title: TQB2916 Injection Combined With Chemotherapy or Penpulimab Injection in the Treatment of Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2916-AK105-II-01
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2023-10

CONDITIONS: Soft Tissue Sarcoma; Melanoma
MeSH Terms: conditions — Sarcoma; Melanoma | interventions — Doxorubicin; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2916 injection + doxorubicin hydrochloride for injection (Experimental): TQB2916 injection + doxorubicin hydrochloride for injection, 21 days as a treatment cycle.
  Interventions: Drug: TQB2916 injection + doxorubicin hydrochloride for injection
- TQB2916 injection+penpulimab injection (Experimental): TQB2916 injection+penpulimab injection , 21 days as a treatment cycle.
  Interventions: Drug: TQB2916 injection+penpulimab injection

INTERVENTIONS:
Drug: TQB2916 injection + doxorubicin hydrochloride for injection — TQB2916 is a humanized immune gamma globulins 2 (IgG2) monoclonal antibody targeting CD40.
  The mechanism of action of doxorubicin is mainly to destroy the DNA structure of tumor cells, thereby killing malignant tumors. It interferes with the DNA synthesis process of cancer cells by targeting DNA and inhibiting enzymes in DNA replication and repair. In addition, doxorubicin can also trigger cross-link breaks in DNA, leading to apoptosis of cancer cells.
  Arms: TQB2916 injection + doxorubicin hydrochloride for injection
Drug: TQB2916 injection+penpulimab injection — TQB2916 is a humanized IgG2 monoclonal antibody targeting CD40. Penpulimab injection is a programmed cell death protein 1 (PD-1) immune checkpoint inhibitor.
  Arms: TQB2916 injection+penpulimab injection

SUMMARY:
This project is a clinical trial on the efficacy and safety of TQB2916 injection combined with chemotherapy or penpulimab injection in solid tumors. This project is divided into two cohorts. Cohort 1 aims to explore the safety and efficacy of specific subtypes of soft tissue sarcoma in subjects; Cohort 2 aims to explore safety and efficacy in subjects with undifferentiated pleomorphic sarcoma and melanoma. A total of 54 subjects are planned to be enrolled in this project.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined this study, signed an informed consent form, and had good compliance.
2. Age: 18-75 years old; Eastern Cooperative Oncology Group Performance Status (ECOG PS) score: 0-1 points; The expected survival period exceeds 3 months.
3. Patients with locally advanced or unresponsive relapsed/metastatic soft tissue sarcoma and melanoma diagnosed by pathology and unable or refused surgery. Cohort 1contains the following subtypes: "dedifferentiated liposarcoma, highly differentiated liposarcoma with dedifferentiated components, leiomyosarcoma (excluding uterine leiomyosarcoma)", and cohort 2 contains undifferentiated pleomorphic sarcoma and melanoma.
4. Cohort 1: No previous history of failure of anthracycline-based chemotherapy. Cohort 2: Previously treated with standard of care.
5. Cohort 2: Previously treated.
6. According to RECIST 1.1 standard, it is confirmed that there is at least one measurable lesion.
7. The main organs are functioning well.
8. Female participants of childbearing age should agree to use contraceptive measures during the study period and within 6 months after the end of the study; Within 7 days prior to enrollment, the serum pregnancy test was negative and must be a non lactating subject; Male participants should agree to use contraceptive measures during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

1. Concomitant diseases and medical history:

   1. Has experienced or currently suffers from other malignant tumors within 5 years.
   2. Unresolved toxic reactions above CommonTerminology Criteria for Adverse Events level 1 caused by any previous treatment;
   3. The research treatment began with significant surgical treatment, open biopsy, or obvious traumatic injury;
   4. Long term unhealed wounds or fractures;
   5. Arterial/venous thrombotic events that have occurred within 6 months and affect current normal function;
   6. Individuals with a history of psychiatric drug abuse who are unable to quit or have mental disorders;
   7. Individuals who have previously undergone splenectomy or received splenic radiotherapy within 3 months prior to enrollment;
   8. Currently present with congenital hemorrhagic or coagulation diseases, or currently undergoing treatment with warfarin;
   9. Subjects with any severe and/or uncontrolled diseases, including:

      * Blood pressure control is still not ideal after dual drug treatment;
      * Suffering from ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia; ≥ Grade 2 unstable angina pectoris;
      * Active or uncontrolled severe infection or unexplained fever>38.5 °C;
      * Cirrhosis and active hepatitis *;
      * Active syphilis patients;
      * Renal failure requiring hemodialysis or peritoneal dialysis;
      * Have a history of immunodeficiency;
      * Poor control of diabetes;
      * Urinary routine indicates urine protein ≥++;
      * Individuals with epilepsy who require treatment;
      * Weight<40 kg and BMI<18.5 kg/m2, or weight loss of ≥ 10% within 3 months.
2. Tumor related symptoms and treatment:

   1. Has received surgery, chemotherapy, radiation therapy, or other anti-cancer therapies before the start of the research treatment;
   2. Before the start of the study treatment, he received the treatment of traditional Chinese patent medicines and simple preparations with anti-tumor indications specified in the National MedicalProducts Administration (NMPA) approved drug directions;
   3. Cohort 1: Previously used doxorubicin exceeding 200mg/m2;
   4. Cohort 2: Undifferentiated multidirectional sarcoma that has previously received more than 2 types of anti vascular tyrosine kinase inhibitors (TKIs), or has previously received relevant immunotherapy drugs;
   5. Previously received antibodies or fusion proteins targeting CD40;
   6. Imaging shows that the tumor invades large blood vessels or has unclear boundaries with large blood vessels, or the researcher determines that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during subsequent studies;
   7. Uncontrollable pleural effusion, pericardial effusion, or ascites that still require repeated drainage;
   8. Severe bone damage caused by tumor bone metastasis may occur in the presence or after enrollment;
   9. Uncontrollable pain related to tumor bone metastasis;
   10. There was central nervous system metastasis before enrollment.
3. Research and treatment related:

   1. History of live attenuated vaccine administration before the start of research treatment or planned live attenuated vaccine administration during the study period;
   2. There is a clear bleeding tendency or clinically significant bleeding symptoms before the first use of medication;
   3. Individuals who have experienced severe hypersensitivity reactions after using monoclonal antibodies, or who are allergic to known components of the investigational drug;
   4. Active autoimmune diseases that require systemic treatment have occurred within 2 years prior to the start of the research treatment.
   5. Diagnosed with immunodeficiency or undergoing systemic glucocorticoid therapy or any other form of immunosuppressive therapy.
4. Participated in clinical trials of other anti-tumor drugs within the first 4 weeks of grouping.
5. According to the researcher's judgment, there are individuals with accompanying diseases that seriously endanger the safety of the subjects or affect the completion of the study, or individuals who are deemed unsuitable for enrollment due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 48 weeks
  Objective response rate refers to the percentage of complete response (CR) or partial response (PR) subjects determined by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or modified RECIST 1.1 for immune based therapeutics(guidelines for response criteria for use in trials testing Immunotherapeutics（iRECIST)) (CR and PR) under iRECIST criteria can occur after imaging disease progression).
Progression-Free Survival (PFS) | Up to 48 weeks
  PFS will be defined as median number of months from the date of randomization until the first documented sign of disease progression or death due to any causes, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 2 years
  Overall survival defined as the time from enrollment to death from any cause.
Duration of Response (DOR) | Up to 48 weeks
  DOR will be defined as median number of months from date of first documented objective response until first documented sign of disease progression or death due to any causes.

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Medical University Affiliated Cancer Hospital, Ürümqi, Xinjiang
  - Zhe Jiang Cancer Hospital, Hangzhou, Zhejiang